CLINICAL TRIAL: NCT02171689
Title: Metabolism and Pharmacokinetics of [14C]- BIBW 2992 MA2 After Administration of Single Doses of 15 mg [14C]- BIBW 2992 MA2 Oral Solution in Healthy Male Volunteers
Brief Title: Metabolism and Pharmacokinetics of [14C]- BIBW 2992 MA2 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.25
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (1):
- BIBW 2992 MA2 (Experimental)
  Interventions: Drug: [14C]- BIBW 2992 MA2

INTERVENTIONS:
Drug: [14C]- BIBW 2992 MA2

SUMMARY:
The aim of the study was to investigate the metabolism and pharmacokinetics of BIBW 2992 MA2 after a single oral dose of [14C]-radiolabelled BIBW 2992 MA2 in healthy male volunteers. Metabolites in human plasma and excretions were measured, the structures of the metabolites analysed and compared with metabolites in animals. In addition, the mass-balance of excretion, the protein binding of [14C]-radioactivity, the plasma concentrations of BIBW 2992 MA2, and the [14C]-radioactivity in blood cells, plasma, urine and faeces were measured. The safety and tolerability of BIBW 2992 were also investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice and local legislation
* Age ≥35 and ≤60 years
* Body Mass Index ≥18.5 kg/m2 and ≤29.9 kg/m2

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of any major surgery within the last four weeks before participation in this study or any bone fracture within the last two months
* History of orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Planned use of any drugs which might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the reference range, unless considered to lack clinical reference
* Male subjects must agree to minimize the risk of female partners becoming pregnant from the dosing day until 3 months after the completion of the study. Acceptable methods of contraception for male volunteers include a vasectomy no less than 3 months prior to dosing, barrier contraception or a medically accepted contraceptive method. For female partners of male volunteers, acceptable methods of contraception include intra-uterine device, tubal ligation, hormonal contraceptive since at least two months and diaphragm with spermicide

Ages: 35 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2006-07; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
[14C]-radioactivity in plasma and whole blood (CBlood cells/Cplasma ratio of [14C]-radioactivity) | up to 96 hours after drug administration
[14C]-radioactivity in urine and faeces (excretion mass balance) | up to 120 hours after drug administration
Measurement of the plasma protein binding of total [14C]-radioactivity | up to 96 hours after drug administration
Concentrations of the analyte in plasma, urine, and faeces | up to 96 hours after drug administration
Cmax (maximum observed concentration of the analyte in plasma) | up to 96 hours after drug administration
tmax (time from dosing to peak concentration (Cmax)) | up to 96 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 96 hours after drug administration
λz (terminal rate constant of the analyte in plasma) | up to 96 hours after drug administration
AUC (area under the concentration-time curve of the analyte in plasma) for different time points | up to 96 hours after drug administration
MRTpo (mean residence time of the analyte molecules in the body after oral administration) | up to 96 hours after drug administration
CL/F (total clearance of the analyte in plasma following extravascular administration) | up to 96 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase following extravascular administration) | up to 96 hours after drug administration
fe0-tz (fraction of analyte eliminated in urine or faeces from 0 to the limit of the last quantifiable data point) | up to 120 hours after drug administration
Aet0-tz (amount of analyte eliminated in urine or faeces from 0 the limit of the last quantifiable data point) | up to 120 hours after drug administration
Plasma concentration time profiles of the analyte | up to 96 hours after drug administration
Plasma concentration-time profiles of total radioactivity in whole blood and plasma | up to 96 hours after drug administration
[14C]-metabolic profile and identification of metabolites in urine, faeces, blood cells and plasma | up to 120 hours after drug administration

SECONDARY OUTCOMES:
Number of patients with clinically relevant changes in vital signs (Pulse rate (PR), systolic and diastolic blood pressure (BP)) | Baseline, day 2, within 14 days after study drug administration
Number of patients with clinically relevant changes in ECG (electrocardiogram) | Baseline, day 2, within 14 days after study drug administration
Number of patients with clinically relevant changes in laboratory parameters | Baseline, day 2, within 14 days after study drug administration
Number of patients with adverse events | up to 27 days
Assessment of tolerability on a 4-point scale | within 14 days after study drug administration